CLINICAL TRIAL: NCT02368743
Title: QUality of Life in pAtients With Mild to modeRate Active procTitis Treated by mesalaZine (Pentasa®)
Acronym: QUARTZ
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 000179
Record Dates: First submitted 2015-02-16; First posted 2015-02-23 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Distal Ulcerative Colitis
MeSH Terms: interventions — Mesalamine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- mesalazine: Treatment according to standard clinical practice.
  Interventions: Drug: mesalazine

INTERVENTIONS:
Drug: mesalazine
  Other Names: Pentasa®

SUMMARY:
This national, observational and multicentre study aims at establishing a picture of real clinical practices management among patients treated with Pentasa®, according to the current therapeutic strategy in proctitis or distal proctosigmoiditis. This study should be able to provide data on patients' health related quality of life, compliance and efficacy in real clinical practice

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older.
* Patient suffering from mild to moderate active proctitis or distal proctosigmoiditis (MAYO score ≥ 3 and ≤ 10) at inclusion based on clinical and endoscopic findings within 6 months before study inclusion.
* Patient with evidence of endoscopic active proctitis or distal proctosigmoiditis (Montreal classification E1 or E2 defined by an involvement not exceeding 25 cm from the anal margin) within 6 months before study inclusion.
* Treatment of the current flare with Pentasa® to induce a remission initiated by the patient, the general practitioner or the gastroenterologist, during the inclusion visit or during the week before the inclusion visit.
* Patient having received oral and written information on the study, without any objections for the use of his/her personal data, and having signed a written Informed Consent Form.

Exclusion Criteria:

* Patient included in an interventional study assessing treatment for active proctitis or distal proctosigmoiditis.
* Patient with left sided, colitis or pancolitis.
* Patient with severe proctitis (MAYO score ≥ 11 at inclusion).
* Patient previously treated with biologics.
* Patient treated with immunosuppressive within 1 month before study inclusion.
* Patient treated with corticosteroids within 2 weeks before study inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Gastroenterologists with private and/or hospital practice
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2018-01-02 (Actual)

PRIMARY OUTCOMES:
Change in Short Inflammatory Bowel Disease Questionnaire (SIBDQ) total score | From baseline to week 8

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (1):
- Gastro-Entérologie et Hépatologie - CHU Brabois (there may be other sites in this country), Vandœuvre-lès-Nancy, France

REFERENCES:
- [Derived] Paupard T, Gonzalez F, Caron B, Siproudhis L, Peyrin-Biroulet L. Real-world evidence of quality of life improvement in patients with distal ulcerative colitis treated by mesalazine: the Quartz study. Eur J Gastroenterol Hepatol. 2022 Dec 1;34(12):1203-1209. doi: 10.1097/MEG.0000000000002444. Epub 2022 Sep 12. PMID 36165055